CLINICAL TRIAL: NCT07055321
Title: A Phase 1, First-in-human, Randomized, Participant- and Investigator-blinded, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Doses of ETH47 in Healthy Participants
Brief Title: A Phase 1, First-in-human Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Doses of ETH47 in Healthy Participants
Acronym: ETH47-101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ethris GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ETH47-101; ISRCTN15391202 (Other: ISRCTN)
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Part A-1 (Experimental)
  Interventions: Drug: ETH47
- Part A-2 (Experimental)
  Interventions: Drug: ETH47
- Part A-3 (Experimental)
  Interventions: Drug: ETH47
- Part A-4 (Experimental)
  Interventions: Drug: ETH47
- Part A-5 (Experimental)
  Interventions: Drug: ETH47
- Part B-1 (Experimental)
  Interventions: Drug: ETH47
- Part B-2 (Experimental)
  Interventions: Drug: ETH47
- Part B-3 (Experimental)
  Interventions: Drug: ETH47
- Part B-4 (Experimental)
  Interventions: Drug: ETH47

INTERVENTIONS:
Drug: ETH47 — Dose level 1; single intranasal administration
  Arms: Part A-1
Drug: ETH47 — Dose level 2; single intranasal administration
  Arms: Part A-2
Drug: ETH47 — Dose level 3; single intranasal administration
  Arms: Part A-3
Drug: ETH47 — Dose level 4; single intranasal administration
  Arms: Part A-4
Drug: ETH47 — Dose level 5; single intranasal administration
  Arms: Part A-5
Drug: ETH47 — Dose level 1; single inhaled administration
  Arms: Part B-1
Drug: ETH47 — Dose level 2; single inhaled administration
  Arms: Part B-2
Drug: ETH47 — Dose level 3; single inhaled administration
  Arms: Part B-3
Drug: ETH47 — Dose level 4; single inhaled administration
  Arms: Part B-4

SUMMARY:
This first-in-human study is designed to evaluate the safety, tolerability, pharmacokinetics and target engagement of ETH47 in healthy participants following single intranasal and single inhaled administration

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF), restriction handbook and in this protocol.
2. Participants who are overtly healthy, as determined by screening assessments and the Investigator's judgement, aged ≥18 and ≤55 years at the time of obtaining informed consent.
3. Body mass index of 18.5 to 32 kg/m2 (inclusive).
4. Participants must agree to use contraception methods.
5. Parts B only: participants must be able to perform reliable and reproducible pulmonary function tests and meet the following criteria at screening:

   1. Forced expiratory volume in one second (FEV1) ≥80 % predicted by third National Health and Nutrition Examination Survey standards, and
   2. Change in FEV1 and forced vital capacity <200 mL, 15 minutes after 4 puffs of inhaled short-acting beta 2-agonists.

Major Exclusion Criteria:

1. History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, neuropsychiatric, autoimmune, or immunosuppressive disorders which, in the Investigator's judgement, puts the participant at risk due to participation in the trial, may influence the results of the trial, or the subject's ability to participate in the trial.
2. Signs or symptoms of upper or lower respiratory tract infection within 2 weeks of randomisation.
3. Participants who are SARS-CoV-2 positive.
4. Known or positive laboratory results at screening for human immunodeficiency virus (HIV) infection, hepatitis B or hepatitis C.
5. Any malignancy except for the following:

   1. Adequately treated basal cell carcinoma or
   2. History of any other cancer where the disease-free period is ≥5 years.
6. The evidence of any other active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, haematology, blood chemistry, serology, and urinalysis.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events (TEAEs) | From treatment until end of study (d 21)
Number of serious adverse events (SAEs) | From enrollment until end of study (day 21)

CONTACTS AND LOCATIONS:
Locations (1):
- CRO, Merthyr Tydfil, United Kingdom

IPD SHARING:
Plan to Share IPD: No